CLINICAL TRIAL: NCT02499445
Title: Comparisons of Myocardial Injury After Using Different Anesthetics Regimens for Off-pump Coronary Artery Bypass Surgery: Remifentanil-based Versus Sevoflurane-sufentanil Balanced Regimen
Brief Title: Myocardial Injury in Remifentanil-based Versus Sevoflurane-sufentanil Balanced Regimens in OPCAB Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Konkuk University Medical Center (Other)
Responsible Party: Principal Investigator, Tae-Yop Kim, MD PhD, Professor of Anesthesiology, Konkuk University Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: KUH1160004
Record Dates: First submitted 2015-03-05; First posted 2015-07-16 (Estimated); Last update posted 2015-07-16 (Estimated); Status verified 2015-07

CONDITIONS: Ischemic Heart Disease
MeSH Terms: conditions — Myocardial Ischemia | interventions — Remifentanil; Propofol; Sufentanil

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Remifentanil and propofol (Active Comparator): remifentanil (0.75 mcg/kg/min) propofol (TCI effect-site concentration 0.8-1.5 mcg/ml)
  Interventions: Drug: Remifentanil; Drug: propofol
- remifentanil and sevoflurane 1 (Active Comparator): remifentanil (0.75 mcg/kg/min) sevoflurane (end-tidal 0.8 vol%)
  Interventions: Drug: Remifentanil; Drug: sevoflurane 1
- sevoflurane 2 and sufentanil (Active Comparator): sevoflurane (end-tidal 1.2-2.8 vol%)-sufentanil (TCI effect site concentration 0.35-0.75 ng/ml)
  Interventions: Drug: sevoflurane 2; Drug: sufentanil

INTERVENTIONS:
Drug: Remifentanil — administering remifentanil for anesthesia maintenance
  Arms: Remifentanil and propofol; remifentanil and sevoflurane 1
Drug: sevoflurane 1 — administering sevoflurane 1 for anesthesia maintenance
  Arms: remifentanil and sevoflurane 1
Drug: sevoflurane 2 — administering sevoflurane 2 for anesthesia maintenance
  Arms: sevoflurane 2 and sufentanil
Drug: propofol — administering propofol for anesthesia maintenance
  Arms: Remifentanil and propofol
Drug: sufentanil — administering sufentanil for anesthesia maintenance
  Arms: sevoflurane 2 and sufentanil

SUMMARY:
In patients undergoing off-pump coronary artery bypass (OPCAB) surgery with different anesthesia regimens: remifentanil (0.75 mcg/kg/min) and propofol (TCI effect-site concentration 0.8-1.5 mcg/ml) (Group -RP); remifentanil (0.75 mcg/kg/min) and sevoflurane (end-tidal 0.8 vol%) (Group-RS), or sevoflurane (end-tidal 1.2-2.8 vol%)-sufentanil (TCI effect site concentration 0.35-0.75 ng/ml) (Group-SS), intergroup difference in the level of Troponin I (c-TnI) and creatinine kinase subtype-MB is determined before surgery (control), during vascular graft harvesting (harvesting), after completing graft construction (postgrafting), and one day after surgery (postoperative).

DETAILED DESCRIPTION:
To determine the difference of myocardial injury upon using different anesthesia regimens: remifentanil-based regimen versus sevoflurane-sufentanil balanced regimen.

Patients undergoing off-pump coronary artery bypass (OPCAB) surgery are randomly allocated to get remifentanil (0.75 mcg/kg/min) and propofol (TCI effect-site concentration 0.8-1.5 mcg/ml) (Group -RP), remifentanil (0.75 mcg/kg/min) and sevoflurane (end-tidal 0.8 vol%) (Group-RS), or sevoflurane (end-tidal 1.2-2.8 vol%)-sufentanil (TCI effect site concentration0.35-0.75 ng/ml) (Group-SS).

Intergroup difference in the level of Troponin I (c-TnI) and creatine kinase-MB is determined before surgery (control), during vascular graft harvesting (harvesting), after completing graft construction (postgrafting), 1 day after surgery (postoperative).

ELIGIBILITY:
Inclusion Criteria:

* patient undergoing OPCAB surgery
* patient signed written informed consent

Exclusion Criteria:

* patient with Intra-aortic balloon pump
* patient with renal replacement therapy
* patient wants to withdraw the participation to the study

Ages: 19 Years to 72 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2007-11; Primary Completion 2014-10 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
troponin I | one day after surgery
  troponin I for myocardial injury

SECONDARY OUTCOMES:
creatinin kinase-MB | one day after surgery
  creatinine kinase-MB

CONTACTS AND LOCATIONS:
Locations (1):
- Konkuk University Medical Center, Seoul, Seoul, South Korea